CLINICAL TRIAL: NCT00000946
Title: A Phase I Trial to Evaluate the HIV-1 SF-2 Recombinant p24 Subunit Vaccine [Chiron Vaccines] Administered as a Novel Boost in "Prime-Boost" Vaccination Regimens With ALVAC-HIV vCP205 [Pasteur Merieux Connaught] and HIV-1 SF-2 rgp120 in MF59 [Chiron Vaccines]
Brief Title: A Study to Test the Safety of Three Experimental HIV Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 032; 10581 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Drug Evaluation; Drug Therapy, Combination; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: HIV p24/MF59 Vaccine
Biological: ALVAC-HIV MN120TMG (vCP205)
Biological: ALVAC-RG Rabies Glycoprotein (vCP65)
Biological: rgp120/HIV-1 SF-2

SUMMARY:
The purpose of this study is to test three experimental HIV vaccines. This study will look at whether it is safe to give these vaccines together and how the immune system responds to the vaccines.

There are a number of studies being performed to test HIV vaccines. The vaccines that seem to be the most promising are canarypox vaccines, known as ALVAC vaccines. The three experimental HIV vaccines used in this study are called ALVAC-HIV vCP205, HIV-1 SF-2 p24, and HIV-1 SF-2 rgp120. The HIV-1 SF-2 p24 and HIV-1 SF-2 rgp120 vaccines are mixed with an adjuvant, which is a substance that increases immune response.

DETAILED DESCRIPTION:
There are currently several Phase I and II clinical trials being performed within AVEG to evaluate different HIV-1 vaccine candidates. The HIV-1 vaccination approach that is furthest along the clinical development pathway is the so-called prime-boost regimen of live recombinant canarypox priming (ALVAC-HIV vCP205) with recombinant subunit protein boosting (HIV-1 SF-2 rgp120 in MF59 adjuvant). The protein boost enhances neutralizing antibody responses against laboratory strains of HIV-1 in assays performed in vitro, as well as enhancing CD4 cell response and increasing the frequency of CD8 cytotoxic T lymphocytes (CTLs). In all of the ALVAC-HIV trials of the prime-boost regimen completed to date, the protein boost has been the HIV-1 SF-2 rgp120 subunit protein. This study is designed to explore whether boosting of live recombinant canarypox vaccination with a novel protein subunit, recombinant HIV-1 SF-2 p24, can enhance the CD4 and CD8 cell responses directed against HIV-1 antigens.

Volunteers are randomized to 1 of 5 groups. All volunteers receive a total of 4 immunizations, administered at Months 0, 1, 3, and 6. Each group receives a different combination of vaccines as follows:

Group 1: ALVAC-HIV vCP205 plus HIV-1 SF-2 p24. Group 2: ALVAC-HIV vCP205 plus MF59 adjuvant and citrate vehicle (control for HIV-1 SF-2 p24 and HIV-1 SF-2 rgp120) at Months 0 and 1; then ALVAC-HIV vCP205 plus HIV-1 SF-2 p24 at months 3 and 6.

Group 3: ALVAC-HIV vCP205 plus control at Months 0 and 1; then ALVAC-HIV vCP205 plus HIV-1 SF-2 p24 combined with HIV-1 SF-2 rgp120 at Months 3 and 6.

Group 4: ALVAC-HIV vCP205 plus control at Months 0 and 1; then ALVAC-HIV vCP205 plus HIV-1 SF-2 rgp 120 at Months 3 and 6.

Group 5: ALVAC-RG vCP65 (control for ALVAC-HIV vCP205) plus control at Months 0,1,3, and 6.

The study lasts for approximately 18 months; patients receive clinical evaluations to measure vaccine safety at 11 study visits at specified time intervals.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are between the ages of 18 and 60.
* Are HIV-negative.
* Are negative for Hepatitis B.
* Have a normal physical exam.
* Are available for 18 months of follow-up.
* Agree to use an effective method of birth control for 1 month before receiving a vaccine and during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of an immunodeficiency, chronic illness, or cancer.
* Have a medical or psychiatric condition which would make you unable to comply with the study.
* Are at higher-risk for HIV infection; for example, have a history of injection drug use in the past year or practice higher risk sexual behavior.
* Have syphilis or tuberculosis.
* Have received a live vaccine in the past 60 days, have ever received an HIV vaccine or placebo in a previous HIV vaccine study, or have ever received a rabies vaccine.
* Have a history of a serious allergic reaction to a vaccine or to any other substance, including neomycin or egg products.
* Have received certain medications.
* Are pregnant or breast-feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Mulligan, MD, Study Chair — Univ of Alabama at Birmingham
Locations (7):
- United States (7):
  - UAB AVEG, Birmingham, Alabama
  - JHU AVEG, Baltimore, Maryland
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - FHCRC/UW Vaccine CRS, Seattle, Washington
  - UW - Seattle AVEG, Seattle, Washington